CLINICAL TRIAL: NCT03024190
Title: The Clinical Effect and Sonographic Findings of Kinesiotaping Combined With Therapeutic Exercise in Upper Extremity Spasticity and Function in Subacute Stroke Patients
Brief Title: Kinesiotaping Combined With Therapeutic Exercise in Upper Extremity Spasticity and Function in Subacute Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CMRPG8F1101
Record Dates: First submitted 2016-12-27; First posted 2017-01-18 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2016-12

CONDITIONS: Stroke; Upper Extremity Spasticity
Keywords: stroke; spasticity; Kinesiotaping; sonography; exercise
MeSH Terms: conditions — Stroke; Muscle Spasticity; Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- with Kinesiotaping (Experimental): * stretching exercises combined with Kinesiotaping
  * regular OT rehabilitation program for 3 weeks
  Interventions: Other: Kinesiotaping; Other: stretching exercise; Other: OT rehabilitation program
- control group (Other): * the patients will receive 15-min stretching exercises
  * regular OT rehabilitation program for 3 weeks
  Interventions: Other: stretching exercise; Other: OT rehabilitation program

INTERVENTIONS:
Other: Kinesiotaping — The technique of Kinesiotaping for spastic wrists and fingers in stroke patients is performed from the proximal interphalangeal joints of all fingers acted on the extensor carpal and digital muscle groups, with an anchor at the proximal one-third forearm.
  Arms: with Kinesiotaping
Other: stretching exercise — 15- min stretching exercise for upper extremity twice daily
Other: OT rehabilitation program — regular rehabilitation program for 3 weeks

SUMMARY:
Poststroke spasticity (PSS) is one of the common complications in stroke patients who had a brain injury leading to limbs weakness and impaired coordination between agonist and antagonist contraction. PSS leads some physical impairments and functional deficits. The clinical managements for PSS are stretching and range of motion (ROM) exercises, antispasticity splint, neuromuscular electrical stimulation, oral medications, local injection with phenol or botulism, or surgery. Recently, some investigators tried to use Kinesiotaping (KT) for spasticity management or postural control. They found some benefits in walking ability and upper extremity function facilitation after stroke.

40 subacute stroke patients with hemiplegia would be enrolled in this study. These 40 patients will be randomly divided into the experimental and control groups. In experimental group (n=20), the patients will perform combined KT and 15- min stretching exercise for upper extremity twice daily and regular rehabilitation program for 3 weeks. In the control group (n=20), the patients will perform 15- min stretching exercise for upper extremity twice daily and regular rehabilitation program for 3 weeks. Before intervention, immediately and 2 week post intervention, all patients will receive associated physical examinations, hand function evaluations, and sonography.

DETAILED DESCRIPTION:
In this study, 40 subacute stroke patients (duration is 3~6 months after stroke) with hemiplegia would be enrolled. Each stroke patient is diagnosed by a neurologist according to the history, physical examination, and brain imaging evaluation. These 40 patients would be randomly divided into a experimental or a control group. All patients in the control and experimental groups will both receive regular rehabilitation therapy including occupational therapy (OT) 3 times per week and one hour for one session OT intervention. Additionally, 15- min stretching exercise for upper extremity twice daily will be performed for 3 weeks in this study. KT intervention in the experimental group: The technique of KT for spastic wrist and fingers in stroke patient will be performed from the proximal interphalangeal joints of all fingers acted on the extensor carpal and digital muscle groups, with an anchor at the proximal one-third forearm. The KT will be applied for 5 days one week for 3 weeks.

In this study, all patients in the control and experimental groups will receive the following evaluations before intervention, immediately post intervention, and 2-week after intervention: Physical examinations (modified shworth scale and Tardieu scale), Hand function evaluation (Fugl-Meyer Assessment for upper extremity, box and block test, and Minnesota Manual Dexterity Test), and Musculoskeletal sonography (sonoelastography and shear wave velocity). SPSS software will be used to record and analysis the collecting data. Investigators will analyze and compare the findings of physical examinations, upper extremity function assessments, and musculoskeletal sonography within and between the experimental and control groups before and after interventions.

ELIGIBILITY:
Inclusion Criteria:

* stroke with hemiplegia (duration is 3~6 months after stroke).
* The upper extremity function of participated patients could perform hand grasp and release movements.

Exclusion Criteria:

* age is younger than 18 years or older than 80 years
* previous history of upper extremity tendon or neuromuscular injury
* any other systemic neuromuscular disease
* cognition or language impairment leading to communication difficulty

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment for upper extremity (FMA-UE) for hand function | baseline (before intervention), changes from baseline FMA-UE scores at 3 weeks and 5 weeks.
  A physical therapist will use Fugl-Meyer assessment for upper extremity (FMA-UE) to evaluate patient's hand function and analyze the changes on the score of it from baseline till third week and fifth week.
Modified Ashworth scale for level of spasticity of affected arm | baseline (before intervention), changes from baseline level of spasticity at 3 weeks and 5 weeks.
  A physical therapist will measure the level of spasticity in affected arm by using modified Ashworth scale.

SECONDARY OUTCOMES:
the change from baseline on hemiplegic upper extremity sonography | baseline (before intervention), changes from baseline sonography results at 3 weeks and 5 weeks.
  for the flexor carpal ulnaris (FCU), flexor carpal radialis (FCR), and flexor digitorum superficialis (FDS) muscles.
  The participants will sit upright and put their upper extremities on the bed with elbow flexion in 90 degree and the forearm full supination. The measured levels for evaluating FCR, FCU, and FDS muscles will be recorded at first time and use the same level after intervention for each patient. The SWV will be done in the transverse plane and be performed at the maximal cross-section area of the muscles and repeatedly measured for 7 times for each muscle. The sonoelastography will be applied in the longitudinal plane of the detected muscles at the same level of the SWV.
Brunnstrom motor recovery stage for motor ability | baseline (before intervention), changes from baseline motor recovery stage at 3 weeks and 5 weeks.
  A physical therapist will measure Brunnstrom motor recovery stage and see the improvement of it from baseline till third week and fifth week.
Modified Tardieu scale for level of spasticity of affected arm | baseline (before intervention), changes from baseline level of spasticity at 3 weeks and 5 weeks.
  A physical therapist will measure the level of spasticity in affected arm by using modified Tardieu scale.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Chi Huang, Bachelor, Principal Investigator — Chang Gung Memorial Hospital

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Background] Francisco GE, McGuire JR. Poststroke spasticity management. Stroke. 2012 Nov;43(11):3132-6. doi: 10.1161/STROKEAHA.111.639831. Epub 2012 Sep 13. No abstract available. PMID 22984012
- [Background] Sommerfeld DK, Eek EU, Svensson AK, Holmqvist LW, von Arbin MH. Spasticity after stroke: its occurrence and association with motor impairments and activity limitations. Stroke. 2004 Jan;35(1):134-9. doi: 10.1161/01.STR.0000105386.05173.5E. Epub 2003 Dec 18. PMID 14684785
- [Background] Ferro JA, Macari M, Eizirik DL. Cold-acclimation improves cold-tolerance of diabetic rats. Comp Biochem Physiol A Comp Physiol. 1987;88(3):425-9. doi: 10.1016/0300-9629(87)90057-0. PMID 2892615
- [Background] Thibaut A, Chatelle C, Ziegler E, Bruno MA, Laureys S, Gosseries O. Spasticity after stroke: physiology, assessment and treatment. Brain Inj. 2013;27(10):1093-105. doi: 10.3109/02699052.2013.804202. Epub 2013 Jul 25. PMID 23885710
- [Background] Watanabe T. The role of therapy in spasticity management. Am J Phys Med Rehabil. 2004 Oct;83(10 Suppl):S45-9. doi: 10.1097/01.phm.0000141130.58285.da. PMID 15448577
- [Background] Bovend'Eerdt TJ, Newman M, Barker K, Dawes H, Minelli C, Wade DT. The effects of stretching in spasticity: a systematic review. Arch Phys Med Rehabil. 2008 Jul;89(7):1395-406. doi: 10.1016/j.apmr.2008.02.015. Epub 2008 Jun 13. PMID 18534551
- [Background] Harvey L, Herbert R, Crosbie J. Does stretching induce lasting increases in joint ROM? A systematic review. Physiother Res Int. 2002;7(1):1-13. doi: 10.1002/pri.236. PMID 11992980
- [Background] Neuhaus BE, Ascher ER, Coullon BA, Donohue MV, Einbond A, Glover JM, Goldberg SR, Takai VL. A survey of rationales for and against hand splinting in hemiplegia. Am J Occup Ther. 1981 Feb;35(2):83-90. doi: 10.5014/ajot.35.2.83. PMID 7223829
- [Background] Basaran A, Emre U, Karadavut KI, Balbaloglu O, Bulmus N. Hand splinting for poststroke spasticity: a randomized controlled trial. Top Stroke Rehabil. 2012 Jul-Aug;19(4):329-37. doi: 10.1310/tsr1904-329. PMID 22750962
- [Background] Mesci N, Ozdemir F, Kabayel DD, Tokuc B. The effects of neuromuscular electrical stimulation on clinical improvement in hemiplegic lower extremity rehabilitation in chronic stroke: a single-blind, randomised, controlled trial. Disabil Rehabil. 2009;31(24):2047-54. doi: 10.3109/09638280902893626. PMID 19874084
- [Background] Walker JB. Modulation of spasticity: prolonged suppression of a spinal reflex by electrical stimulation. Science. 1982 Apr 9;216(4542):203-4. doi: 10.1126/science.7063882.
- [Background] Ring H, Weingarden H. Neuromodulation by functional electrical stimulation (FES) of limb paralysis after stroke. Acta Neurochir Suppl. 2007;97(Pt 1):375-80. doi: 10.1007/978-3-211-33079-1_49. PMID 17691399
- [Background] Lin Z, Yan T. Long-term effectiveness of neuromuscular electrical stimulation for promoting motor recovery of the upper extremity after stroke. J Rehabil Med. 2011 May;43(6):506-10. doi: 10.2340/16501977-0807. PMID 21533330
- [Background] Sahin N, Ugurlu H, Albayrak I. The efficacy of electrical stimulation in reducing the post-stroke spasticity: a randomized controlled study. Disabil Rehabil. 2012;34(2):151-6. doi: 10.3109/09638288.2011.593679. Epub 2011 Oct 15. PMID 21999668
- [Background] Yan T, Hui-Chan CW. Transcutaneous electrical stimulation on acupuncture points improves muscle function in subjects after acute stroke: a randomized controlled trial. J Rehabil Med. 2009 Apr;41(5):312-6. doi: 10.2340/16501977-0325. PMID 19363561
- [Background] Goldstein EM. Spasticity management: an overview. J Child Neurol. 2001 Jan;16(1):16-23. doi: 10.1177/088307380101600104. PMID 11225951
- [Background] Wagstaff AJ, Bryson HM. Tizanidine. A review of its pharmacology, clinical efficacy and tolerability in the management of spasticity associated with cerebral and spinal disorders. Drugs. 1997 Mar;53(3):435-52. doi: 10.2165/00003495-199753030-00007. PMID 9074844
- [Background] Olvey EL, Armstrong EP, Grizzle AJ. Contemporary pharmacologic treatments for spasticity of the upper limb after stroke: a systematic review. Clin Ther. 2010 Dec;32(14):2282-303. doi: 10.1016/j.clinthera.2011.01.005. PMID 21353101
- [Background] Bakheit AM, Thilmann AF, Ward AB, Poewe W, Wissel J, Muller J, Benecke R, Collin C, Muller F, Ward CD, Neumann C. A randomized, double-blind, placebo-controlled, dose-ranging study to compare the efficacy and safety of three doses of botulinum toxin type A (Dysport) with placebo in upper limb spasticity after stroke. Stroke. 2000 Oct;31(10):2402-6. doi: 10.1161/01.str.31.10.2402. PMID 11022071
- [Background] McCrory P, Turner-Stokes L, Baguley IJ, De Graaff S, Katrak P, Sandanam J, Davies L, Munns M, Hughes A. Botulinum toxin A for treatment of upper limb spasticity following stroke: a multi-centre randomized placebo-controlled study of the effects on quality of life and other person-centred outcomes. J Rehabil Med. 2009 Jun;41(7):536-44. doi: 10.2340/16501977-0366. PMID 19543664
- [Background] Ashby J. Choice of route of exposure in mammalian genotoxicity experiments. Environ Mol Mutagen. 1987;10(4):439-40. doi: 10.1002/em.2850100414. No abstract available. PMID 3678211
- [Background] Lin YC. Botulinum toxin injection for post-stroke spasticity. Muscle Nerve. 2014 Jun;49(6):932. doi: 10.1002/mus.24216. Epub 2014 Apr 8. No abstract available. PMID 24639239
- [Background] Phadke CP, Ismail F, Boulias C, Gage W, Mochizuki G. The impact of post-stroke spasticity and botulinum toxin on standing balance: a systematic review. Expert Rev Neurother. 2014 Mar;14(3):319-27. doi: 10.1586/14737175.2014.887443. Epub 2014 Feb 10. PMID 24506569
- [Background] Rojhani-Shirazi Z, Amirian S, Meftahi N. Effects of Ankle Kinesio Taping on Postural Control in Stroke Patients. J Stroke Cerebrovasc Dis. 2015 Nov;24(11):2565-71. doi: 10.1016/j.jstrokecerebrovasdis.2015.07.008. Epub 2015 Aug 29. PMID 26321149
- [Background] Boeskov B, Carver LT, von Essen-Leise A, Henriksen M. Kinesthetic taping improves walking function in patients with stroke: a pilot cohort study. Top Stroke Rehabil. 2014 Nov-Dec;21(6):495-501. doi: 10.1310/tsr2106-495. PMID 25467397
- [Background] Janda R, Cencora A, Uzieblo W. [Lysis of thrombi and emboli by means of streptokinase. I. Activation of fibrinolysis, mechanism of plasmin activity, indications and contra-indications, treatment principles]. Przegl Lek. 1969;25(10):701-5. No abstract available. Polish. PMID 4242965
- [Background] Jaraczewska E, Long C. Kinesio taping in stroke: improving functional use of the upper extremity in hemiplegia. Top Stroke Rehabil. 2006 Summer;13(3):31-42. doi: 10.1310/33KA-XYE3-QWJB-WGT6. PMID 16987790
- [Background] Hamesh Dash DM. Florence Nightingale's writings. Nurs J India. 1972 May;63(5):149 passim. No abstract available. PMID 4483417
- [Background] Pandyan AD, Johnson GR, Price CI, Curless RH, Barnes MP, Rodgers H. A review of the properties and limitations of the Ashworth and modified Ashworth Scales as measures of spasticity. Clin Rehabil. 1999 Oct;13(5):373-83. doi: 10.1191/026921599677595404. PMID 10498344
- [Background] Haugh AB, Pandyan AD, Johnson GR. A systematic review of the Tardieu Scale for the measurement of spasticity. Disabil Rehabil. 2006 Aug 15;28(15):899-907. doi: 10.1080/09638280500404305. PMID 16861197
- [Background] Li F, Wu Y, Li X. Test-retest reliability and inter-rater reliability of the Modified Tardieu Scale and the Modified Ashworth Scale in hemiplegic patients with stroke. Eur J Phys Rehabil Med. 2014 Feb;50(1):9-15. Epub 2013 Dec 5. PMID 24309501
- [Background] van Rijthoven AW, Dijkmans BA, Goei The HS, Hermans J, Montnor-Beckers ZL, Jacobs PC, Cats A. Cyclosporin treatment for rheumatoid arthritis: a placebo controlled, double blind, multicentre study. Ann Rheum Dis. 1986 Sep;45(9):726-31. doi: 10.1136/ard.45.9.726. PMID 3532966
- [Background] Ansari NN, Naghdi S, Hasson S, Azarsa MH, Azarnia S. The Modified Tardieu Scale for the measurement of elbow flexor spasticity in adult patients with hemiplegia. Brain Inj. 2008 Dec;22(13-14):1007-12. doi: 10.1080/02699050802530557. PMID 19117179
- [Background] Kesikburun S, Yasar E, Adiguzel E, Guzelkucuk U, Alaca R, Tan AK. Assessment of Spasticity With Sonoelastography Following Stroke: A Feasibility Study. PM R. 2015 Dec;7(12):1254-1260. doi: 10.1016/j.pmrj.2015.05.019. Epub 2015 May 30. PMID 26032348
- [Background] Park GY, Kwon DR. Sonoelastographic evaluation of medial gastrocnemius muscles intrinsic stiffness after rehabilitation therapy with botulinum toxin a injection in spastic cerebral palsy. Arch Phys Med Rehabil. 2012 Nov;93(11):2085-9. doi: 10.1016/j.apmr.2012.06.024. Epub 2012 Jul 7. PMID 22776155